CLINICAL TRIAL: NCT00988169
Title: A Phase II Trial of Erlotinib and AT-101 in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients With EGFR Activating Mutations
Brief Title: Erlotinib and AT-101 in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients With Epidermal Growth Factor Receptor (EGFR) Activating Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ascenta Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-026
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: AT-101; erlotinib; Unresectable Stage IIIB; 09-026
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

ARMS (1):
- oral erlotinib and pulsed doses of oral AT-101 (Experimental): This will be an open-label, single institution, phase II trial. The study will assess the efficacy of the combination of the epidermal growth factor receptor tyrosine kinase inhibitor, erlotinib, and the novel pan-Bcl-2 inhibitor, AT-101, in treatment-naïve advanced (Wet Stage IIIB and IV)NSCLC patients with EGFR activating mutations A planned pause of 21 days will be performed after enrollment of the 10th and 20th patient to assess for excessive toxicity.
  Interventions: Drug: oral erlotinib and pulsed doses of oral AT-101

INTERVENTIONS:
Drug: oral erlotinib and pulsed doses of oral AT-101 — Patients will receive oral erlotinib 100 mg daily and pulsed doses of oral AT-101 given 40 mg twice daily on days 1-3 of a 21-day cycle. If the initial combination of erlotinib and AT-101 is tolerated, dose escalation of erlotinib to 150 mg daily will be allowed at the discretion of the treating investigator at the start of cycle 2. Patients will continue receiving treatment on study until they refuse further therapy, develop evidence of progressive disease, or develop unacceptable toxicity or a medical condition that would, in the judgment of the investigator,

SUMMARY:
Advanced stage lung cancer is generally treated with anti-cancer medication called chemotherapy. Most lung cancer is caused by cigarette smoking. However, some lung cancers develop in people who never smoked or who only smoked for a short period of time. This type of lung cancer may respond to a medication called erlotinib (Tarceva). Erlotinib is an anticancer pill that is approved by the Food and Drug Administration (FDA) for use in patients with advanced lung cancer. Unfortunately, erlotinib does not work for all patients or only works for a period of time. The doctors are trying to find ways to improve the effect of erlotinib by combining it with another anti-cancer medication.

Ascenta Therapeutics, Inc. has developed a drug called AT-101 as a potential treatment for cancer. AT-101 is an investigational drug. That means that AT-101 is not approved by the United States Food and Drug Administration (FDA) for general use. The FDA does permit its use in studies like this one to determine whether it is safe and effective.

This is the first study to examine the effects of AT-101 and erlotinib. It is hoped that by combining AT-101 with erlotinib, AT-101 may help erlotinib work better to shrink lung cancer. Studies that have been performed in the laboratory suggest that AT-101 in combination with erlotinib may be more effective at shrinking tumors than erlotinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent form; the consent form must be signed by the patient prior to any study-specific procedures.
* Patients age ≥ 18 years with histologically confirmed wet Stage IIIB (with malignant pleural effusion) or Stage IV non-small cell lung cancer (metastatic or recurrent).
* Pathologic confirmation of non-small cell lung cancer at Memorial Sloan-Kettering Cancer Center.
* Presence of exon 19 or exon 21 EGFR activating mutation.
* No prior EGFR tyrosine kinase therapy.
* No prior systemic therapy for advanced NSCLC (Stage IIIB with malignant effusion or Stage IV)
* Karnofsky performance status > or = to 70% OR ECOG performance status ≤ 2.
* Measurable disease defined as greater than or equal to one known/suspected malignant lesion > or = to 1 cm measurable in two dimensions.
* Adequate hematologic, renal, and/or hepatic function: WBC > or = to 3,000/ul, hemoglobin > or = to 9.0 g/dl, platelet count > or = to 100,000/ul, total bilirubin ≤ 1.5 X UNL, AST ≤ 2.5 X UNL, and serum creatinine within 1.5 x the upper limit of normal (<1.95 at MSKCC) or calculated creatinine clearance > or = to 60 ml/min.
* Able to swallow and retain oral medication.
* Willingness and ability to comply with study procedures and follow-up examination.
* Four weeks since any major surgery, completion of radiation, or completion of all prior chemotherapy.
* Acute toxicities of any prior therapy must have resolved to < Grade 1 or baseline prior to starting study therapy.
* Effective contraception.

Exclusion Criteria:

* Prior treatment with gefitinib, erlotinib, or other EGFR tyrosine kinase inhibitor therapy.
* Concurrent cytotoxic or biological therapy.
* Known KRAS mutation.
* History within the past 6 months of myocardial infarction, cardiac stent placement, or intermittent ischemia with troponin leak.
* Active secondary malignancy or history of other malignancy within the last 3 years except non-melanoma skin cancer and in-situ carcinoma of the cervix.
* Active, serious comorbid medical conditions including severe infection, malnutrition, unstable angina, congestive heart failure (New York Heart Association Class III or IV), pulmonary fibrosis, or condition that would be felt by treating physician to preclude safe participation in the clinical trial.
* Patients with malabsorption syndrome or diseases significantly affecting the gastrointestinal tract including prior gastric resection or small bowel resection, inflammatory bowel disease, or partial or complete small bowel obstruction.
* Unstable brain or leptomeningeal metastases including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Women who are pregnant or breast-feeding.
* Inability/unwillingness to comply with protocol treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Erlotinib and Pulsed Doses of Oral AT-101: Treatment-naïve advanced (Wet Stage IIIB and IV)NSCLC patients with EGFR activating mutations.
Period: Overall Study
Arm/Group | Oral Erlotinib and Pulsed Doses of Oral AT-101
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Erlotinib and Pulsed Doses of Oral AT-101
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Objective Response Rate
Description: (CR+PR, by WHO Criteria for Standard Bidimensional Tumor Measurement) After One 21-day Cycle of Combination Therapy With Erlotinib and AT-101
Time Frame: 21 days after cycle one
Measure: Number; unit: participants
Arm/Group | Oral Erlotinib and Pulsed Doses of Oral AT-101
Number analyzed (Participants) | 5
participants
  Minor Response (MR) | 1
  Stable Disease (SD) | 3
  Partial Response (PR) | 1

ADVERSE EVENTS:
Arm/Group | Oral Erlotinib and Pulsed Doses of Oral AT-101
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Erlotinib and Pulsed Doses of Oral AT-101 (N=5)
Hypotension (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Erlotinib and Pulsed Doses of Oral AT-101 (N=5)
ALT, SGPT (Blood and lymphatic system disorders) | 3 (3)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes